CLINICAL TRIAL: NCT07156565
Title: A Seamless Phase 1/2 Open-label Study to Evaluate the Safety, Determine the Maximum Tolerated Dose of Administered Activity, and Evaluate the Efficacy of the Therapeutic Radiopharmaceutical [Ac 225]-RTX-2358 in the Treatment of Relapsed or Refractory Sarcoma
Brief Title: Actinium Therapy for Late-stage Aggressive Sarcomas
Acronym: ATLAS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ratio Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RTX-2358-101
Record Dates: First submitted 2025-01-17; First posted 2025-09-05 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-12

CONDITIONS: Advanced Soft Tissue Sarcoma
Keywords: Radioligand Therapy; Sarcoma; Relapsed or refractory sarcoma; Soft tissue sarcoma; Radiopharmaceuticals; Theranostics; advanced soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Recurrence

STUDY DESIGN:
Intervention Model Description: The Phase 1 portion of the study is a "3+3" dose escalation design planned for 3 cohorts/groups/dose levels
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment with [Ac 225]RTX-2358 (Experimental): The study design is a 3+3 escalating group design.
  Interventions: Drug: [Ac 225]RTX-2358; Diagnostic Test: [Cu64]LNTH-1363S

INTERVENTIONS:
Drug: [Ac 225]RTX-2358 — [Ac225]RTX-2358 will be given as an intravenous injection once every 8 weeks for up to 6 doses. Each group (3 total) will receive a set administered activity level (dose) of [Ac 225]RTX 2358 given once every 8 weeks. The first group will received the lower dose, the second group will received the mid level dose, and the third group the highest dose. A Safety Review Committee will determine when/if it is appropriate to allow the next group to proceed.
Diagnostic Test: [Cu64]LNTH-1363S — [Cu64]LNTH-1363S is a investigational radioactive diagnostic imaging agent to demonstrate that the tumor expresses Fibroblast Activation Protein. An imaging test is performed after a single injection with [Cu64]LNTH-1363S 13-35 days before the first administration of study drug [AC225]RTX-2358 to confirm that the sarcoma has FAP expression.

SUMMARY:
The goal of this clinical trial is to learn about the safety of drug [Ac225]RTX-2358 and the diagnostic imaging agent [Cu64]LNTH-1363S. Additionally Ratio Therapeutics will learn if [Ac225]RTX-2358 drug is effective in treating advanced sarcoma.

The main questions the study aims to answer in Phase/Part 1 of the trial are:

* Is [Ac225]RTX-2358 tolerable or does it cause toxicities (medical problems) in patients.
* What is the most tolerable dose of [Ac225]RTX-2358
* Does the treatment show effectiveness on advanced sarcoma

Participants will:

* Take drug [Ac225]RTX-2358 once every 8 weeks (4 cycle target; 6 cycle maximum) over a period of 12 months
* Visit the clinic three times for the first week of cycle one, then once a week for the remaining 7 weeks of cycle 1 for check-ups and tests.
* For cycles 2-6: patient will visit the clinic once every 2 weeks for checkups and tests
* Remain in long term follow-up for a period of four additional years

DETAILED DESCRIPTION:
RTX-2358-101 is an open-label, seamless, Phase1/2 clinical study to evaluate safety, tolerability, dosimetry, biodistribution, pharmacokinetic (PK), and anti-tumor activity of [Ac225]RTX-2358. [Ac 225]-RTX-2358 for patients with relapsed or treatment-resistant soft tissue sarcoma.

The study consists of two phases, an ascending administered activity phase (Phase1) and an expansion phase (Phase 2). In the Phase 1 portion of the trial patients will be divided into three groups, each group receiving a higher dose than the last. A standard "3 + 3" dose escalation approach will be used, meaning three patients will start in each group, and more may be added if needed, to confirm safety.

Patients must be 18 or older, have soft tissue sarcoma that can be measured by imaging, and meet specific health requirements, including good organ function and a positive PET scan. Each treatment cycle in the phase 1 portion of the study involves a single injection on Day 1, followed by eight weeks of monitoring. Patients have a target of four cycles of treatment, with the possibility of two more (six maximum), if their side effects are mild and their disease hasn't worsened.

A Safety Review Committee (SRC) will review the data from each group in the Phase 1 portion to decide when it's safe to move to the next dose level. Once dose escalation of all cohorts is approved, patients can be added to two higher-dose groups to gather additional safety and preliminary data on effectiveness. Patients that receive at least one treatment in the Phase 1 portion of the study, will be followed for an initial period of 48 weeks for safety. After the first year, patients will have telephone check-ins every six months for up to four more years to track long-term safety, disease progression, and overall survival.

The Phase 2 portion of the study will evaluate the efficacy and safety of [Ac225]RTX-2358 on up to 50 patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* History of relapse and refractory soft tissue sarcoma.

  1. Histological confirmation of sarcoma at any point since diagnosis
  2. At least 1 prior treatment regimen
* Measurable disease as per RECIST (v1.1) for soft tissue sarcoma that is also positive on FAPi PET/CT or PET/MRI scan.

So keep the inclusion criteria bullet, just not include the exact definition of positive scan.

* ECOG performance status of 0 or 1.
* Adequate Organ reserve and renal function as evidenced by:

  1. Neutrophil count ≥ 1200 µL without granulocyte colony stimulating factor
  2. Platelet count ≥ 100,000 µL
  3. Hemoglobin ≥ 8 g/dL
  4. Total bilirubin level ≤ 1.5 × upper limit of normal (ULN).
  5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN.
  6. Calculated creatinine clearance ≥ 60 mL/min. 6. Coagulation parameters (prothrombin time, international normalized ratio and activated partial thromboplastin time) ≤ 1.5 × ULN 7. All patients (males and females of childbearing potential) must agree to practice 2 forms of highly effective contraceptive precautions to prevent pregnancy from the time consent is signed and throughout the trial.

     8. The patient or the patient's legal representative must be willing and able to provide written informed consent.

     Exclusion Criteria:
* History of whole pelvic irradiation.
* History of radioligand therapy.
* Treatment within 14 days prior to first administration with:

  1. Palliative surgery or external beam radiation.
  2. Approved anticancer therapy including chemotherapy or immunotherapy.
  3. Any investigational therapy.
  4. Any major surgery (e.g., requiring general anesthesia).
* Patients who are scheduled for external beam radiation therapy or radioligand therapy during the study period.
* Congestive heart failure > Class II New York Heart Association Functional Classification, current pericarditis, myocardial infarction within 6 months, or symptomatic coronary artery disease.
* Patients with uncontrollable incontinence.
* Unstable or clinically significant concurrent medical condition that would, in the opinion of the Investigator, jeopardize the safety of a patient and/or their compliance with the protocol.
* Active infection requiring systemic antibacterial/antibiotic, antifungal, or antiviral therapy. Chronic antiviral therapy for stable viral disease can be included.
* History of active fibrotic condition.
* Any active malignancy other than sarcoma that requires treatment (.
* Currently pregnant or lactating.
* Known allergy to any of the study drugs or their excipients.- Inability or unwillingness to comply with any of the required imaging studies or study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety (Frequency and severity of treatment emergent adverse events (TEAEs), Dose Limiting Toxicities (DLTs), serious adverse events (SAEs) and adverse events of special interest) of [Ac225-]RTX-2358 | 48 weeks
  Frequency and severity of treatment emergent adverse events (TEAEs), Dose Limiting Toxicities (DLTs), serious adverse events (SAEs) and adverse events of special interest (AESIs).
  Preliminary efficacy response across all cycles in Phase 1.

SECONDARY OUTCOMES:
Determination the normal tissue radiation dosimetry of [Ac225]RTX-2358 | Day 1, 3, 8
  Radiation absorbed dose estimates for selected normal tissues.
  Analysis of radioactive blood samples for select timepoints.
Evaluate the preliminary anti-tumor activity of [Ac225]RTX-2358 in patients with relapsed or refractory soft tissue sarcoma | 48 weeks
  Objective response rate (ORR), defined as the proportion of patient with a complete response (CR) or partial response (PR), per RECISTv1.1.
Evaluate the preliminary anti-tumor activity of [Ac225]RTX-2358 in patients with relapsed or refractory soft tissue sarcoma | 48 weeks
  Duration of Response (DOR), defined as the duration of time from first date of observed response (CR or PR), to first date of disease progression of death from any cause.
Evaluate the safety and tolerability of [Cu-64]LNTH-1363S | Up to 2 weeks after the [Cu64]LNTH-1363S injections
  Frequency and severity of Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAE)s
Determine the pharmacokinetics (PK) of [Ac225]RTX-2358 | Day 1, 3 and 8
  Clearance, area under the concentration time curve over 4 hours (AUC0 4) and to the last measurable concentration (AUC0 last), for [Ac 225]RTX 2358.
Determine the pharmacokinetics (PK) of [Ac225]RTX-2358 | Day 1, 3 and 8
  (Cmax) for [Ac 225]RTX 2358
Determine the pharmacokinetics (PK) of [Ac225]RTX-2358 | Day 1, 3 and 8
  Half life for [Ac 225]RTX 2358
Assess impact of treatment to quality of life (QoL) - European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLC-C30 Version 3) | 48 Weeks
  Change from baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLC-C30 Version 3)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - UCLA, Los Angeles, California
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloane Kettering Cancer Center, New York, New York
  - Case Western, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No